CLINICAL TRIAL: NCT07031596
Title: Study on the Weight Loss Effects and Mechanisms of Probiotic Preparation Intervention in Weight Cyclers: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Study on the Weight Loss Effects and Mechanisms of Probiotic Preparation Intervention in Weight Cyclers
Acronym: Probiotic
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K7816
Record Dates: First submitted 2025-06-04; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Obesity and Obesity-related Medical Conditions
MeSH Terms: conditions — Obesity | interventions — S100 Proteins; Caloric Restriction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Probiotic Group 1 (Experimental): Daily oral administration of Probiotic Formulation 1 (2 bottles, twice daily) for 84 days.
  Interventions: Dietary Supplement: WONDERLAB SHAPE100™ Ready-to-Eat Probiotic Food (S100).
- Probiotic Group 2 (Experimental): Daily oral administration of Probiotic Formulation 2 (2 bottles, twice daily) for 84 days.
  Interventions: Dietary Supplement: WONDERLAB SHAPE100™ Ready-to-Eat Probiotic Food (S100) + WONDERLAB Weight Management Probiotic Food.
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: WONDERLAB SHAPE100™ Ready-to-Eat Probiotic Food (S100). — Product : WONDERLAB SHAPE100™ Ready-to-Eat Probiotic Food (S100). Ingredients : Stachyose, fructooligosaccharides, isomaltooligosaccharides, maltodextrin, Lactiplantibacillus plantarum CECT7527, Lactiplantibacillus plantarum CECT7528, Lactiplantibacillus plantarum CECT7529, Lactobacillus acidophilus GOLDGUT-LA100, and Epigallocatechin gallate (EGCG).
  Administration : Twice daily (2 bottles per dose) after meals for 12 weeks.
  Other Names: Calorie-Restricted Diet
  Arms: Probiotic Group 1
Dietary Supplement: WONDERLAB SHAPE100™ Ready-to-Eat Probiotic Food (S100) + WONDERLAB Weight Management Probiotic Food. — Product : WONDERLAB SHAPE100™ Ready-to-Eat Probiotic Food (S100) + WONDERLAB Weight Management Probiotic Food.
  Ingredients :
  S100 Components : As above. Weight Management Components : Isomaltooligosaccharides, fructooligosaccharides, maltodextrin, Lactobacillus fermentum K7-Lb1, Lactobacillus fermentum K8-Lb1, Lactobacillus fermentum K11-Lb3, Euglena gracilis, and phosphatidylserine.
  Administration : Twice daily (2 bottles per dose) after meals for 12 weeks.
  Other Names: Calorie-Restricted Diet
  Arms: Probiotic Group 2
Dietary Supplement: Placebo — Daily oral administration of maltodextrin-based placebo (identical in taste, appearance, and packaging to probiotic products) twice daily (2 bottles per dose) for 12 weeks.
  Other Names: Calorie-Restricted Diet
  Arms: Placebo

SUMMARY:
1. Study Background and Purpose Obesity is a complex chronic disease closely linked to comorbidities such as cardiovascular disease, hypertension, and diabetes. With lifestyle changes, obesity prevalence continues to rise. Current treatments focus on weight loss through dietary control and exercise, but weight regain is common due to metabolic adaptations (e.g., post-caloric restriction). Gut microbiota play a critical role in weight management, and probiotics may reduce weight regain by modulating appetite and metabolism. Studies suggest probiotics enhance satiety and reduce appetite. This study aims to evaluate the potential of probiotics in obesity management, specifically their impact on gut microbiota modulation and hormonal regulation to mitigate weight regain. Ethical approval has been obtained from the Peking Union Medical College Hospital Ethics Committee.
2. Study Design

   This 198-participant, randomized, interventional trial will assign subjects to three groups (1:1:1 ratio):

   Placebo group (maltodextrin-based placebo) Probiotic Group 1 Probiotic Group 2 Randomization will be conducted via sealed envelopes (no researcher/participant bias). All groups receive standardized nutritional counseling, caloric restriction plans, and body composition assessments. Probiotics (produced by Shenzhen BaoShiJian Biotechnology Co., Ltd., compliant with standard Q/BSJ 0023S-2024) will be administered orally (2 bottles twice daily) for 84 days .
3. Study Procedure Informed Consent : Required before participation. Screening Phase : Demographic history, medical records, concomitant medications, validated questionnaires, body composition analysis, and blood/urine/stool tests.

   Intervention : Daily probiotic or placebo intake for 84 days. Follow-ups : Visits at Day 42 and Day 85 for adherence checks, anthropometric measurements, and repeat testing.
4. Study Completion Duration : 84 days. Post-Study : Placebo group receives 1-month free probiotic supply; others return to standard care. A 30-day post-study follow-up (phone/WeChat) will assess safety.

   Withdrawal : Participants may exit anytime. Investigators may withdraw participants for safety reasons.
5. Potential Benefits Personalized nutrition counseling and body composition reports. Free clinical evaluations and health coaching. Contribution to novel weight management strategies for weight-cycling populations.
6. Risks and Discomforts Adverse Events : Gastrointestinal symptoms or discomfort. Immediate reporting required for medical management.

Inconveniences :

3 on-site visits (blood/urine/stool tests, anthropometry) with fasting blood draws (~7-20 mL/session).

1 telehealth visit (25 min questionnaire). Daily diary cards. Compensation : 150 RMB travel reimbursement + study-provided scales. 7. Alternative Options

Participants may opt for:

Intermittent fasting. Pharmacotherapy (e.g., GLP-1 agonists). Standard dietary recommendations. 8. New Information Any significant findings during the trial will be communicated to participants, who may choose to continue or withdraw.

9. Costs and Reimbursement No-cost : All investigational products (probiotics/placebo), lab tests, and body composition analyses.

Reimbursement : 150 RMB travel compensation + study tools (body fat scale, food scale, tape measure).

10. Adverse Event Policy All injuries attributed to the intervention will be covered by Shenzhen BaoShiJian Biotechnology Co., Ltd. 's insurance. Legal liability extends beyond insurance coverage.

ELIGIBILITY:
Inclusion Criteria:

* Obesity : BMI ≥28 kg/m² and <35 kg/m².
* Weight Cycling History :

Documented weight loss attempts within the past 2 years (≥3 episodes) with ≥5% body weight fluctuation.

* Age : 18-60 years (inclusive), male or female.
* Comprehension and Voluntariness : Ability to understand the weight loss protocol and willingness to complete the full study.
* Informed Consent : Signed informed consent form.

Exclusion Criteria:

* Weight-Loss Medications : Current use of medications affecting weight (e.g., orlistat, GLP-1 receptor agonists, metformin).
* Diabetes Mellitus : Diagnosed diabetes or use of antidiabetic medications.
* Severe Metabolic Abnormalities :

Triglycerides >2.5× upper limit of normal (ULN) Cholesterol >2.5× ULN (method-dependent) Fasting whole-blood glucose >11.1 mmol/L Uric acid >2× ULN

* Pregnancy/Lactation : Currently pregnant, breastfeeding, or planning pregnancy within 3 months.
* Severe Organ Dysfunction : Advanced cardiovascular, hepatic, pulmonary, renal, or other critical organic diseases.
* Thyroid Disorders : Diagnosed hyperthyroidism or hypothyroidism.
* Gastrointestinal Diseases : History of acute/chronic or active gastrointestinal disorders.
* Antibiotic Use : Oral/intravenous antibiotics within the past month.
* Psychiatric Disorders : Severe mental illness requiring routine psychiatric medication.
* Secondary Obesity : Hypothalamic obesity, Cushing's syndrome, hypogonadism-related obesity, etc.
* Specific Diets : Long-term vegan or restrictive dietary patterns.
* Weight Instability : ≥10% body weight change within the past 3 months.
* Compliance Concerns : Poor compliance or inability to adhere to the weight loss protocol (as judged by the investigator).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 198 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with >5% Body Weight Loss | From baseline (D0) to end of intervention (D85 ±7 days)
  Proportion of participants achieving ≥5% reduction in body weight from baseline (D0) to end of intervention (D85).

SECONDARY OUTCOMES:
Change in Power of Food Scale (PFS) Score | From baseline (D0) to end of intervention (D85 ±7 days)
  The PFS assesses hedonic hunger on a 15-75 scale. Higher scores indicate greater responsiveness to the food environment.
Change in Fasting Insulin Concentration | From baseline (D0) to end of intervention (D85 ±7 days)
  Measured in fasting state using immunoassay.Unit of Measure: μU/mL
Change in Body Weight | From baseline (D0) to end of intervention (D85 ±7 days)
  Measured in kilograms using a calibrated digital scale.
Change in Triglyceride Concentration | From baseline (D0) to end of intervention (D85 ±7 days)
  Fasting triglycerides measured via enzymatic assay.Unit of Measure: mmol/L
Change in Gut Microbial α-Diversity (Shannon Index) | From baseline (D0) to end of intervention (D85 ±7 days)
  Microbial α-diversity will be assessed using the Shannon index. Higher values indicate greater microbial diversity.
Number of Participants with Treatment-Related Adverse Events (AEs) | From baseline (D0) to end of intervention (D85 ±7 days)
  adverse events will be recorded and graded using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Change in Dutch Eating Behavior Questionnaire (DEBQ) Score | From baseline (D0) to end of intervention (D85 ±7 days)
  The DEBQ includes three subscales: emotional, external, and restrained eating. Each subscale is scored from 1 (low tendency) to 5 (high tendency). Higher scores indicate a stronger presence of the eating behavior.
Change in Fasting Ghrelin Concentration | D0 to D85 ±7 days
  Active ghrelin measured via ELISA.Unit of Measure: pg/mL
Change in LDL-Cholesterol Concentration | From baseline (D0) to end of intervention (D85 ±7 days)
  LDL-C calculated using Friedewald formula or direct measurement.Unit of Measure: mmol/L
Change in Gastrointestinal Symptom Score | From baseline (D0) to end of intervention (D85 ±7 days)
  GI symptoms including bloating and diarrhea will be rated on a 5-point Likert scale (1 = none, 5 = very severe). Higher scores indicate more severe symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes